CLINICAL TRIAL: NCT04425733
Title: A Study to Assess the Safety, Tolerability, and Pharmacodynamics of Multiple Dose MK-5475 in Participants With Hypoxemia Due to COVID-19 Pneumonia
Brief Title: Frespaciguat (MK-5475) in Participants With Hypoxemia Due to COVID-19 Pneumonia (MK-5475-009)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 5475-009; MK-5475-009 (Other: Merck Protocol Number); 2020-002062-14 (EudraCT Number)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Coronavirus Disease 2019 (COVID-19); Pneumonia; Hypoxemia
MeSH Terms: conditions — COVID-19; Pneumonia; Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Panel A Frespaciguat 180 µg (Experimental): Participants receive 180 µg of frespaciguat once daily (QD) via inhalation from Days 1-7.
  Interventions: Drug: Frespaciguat
- Panel A Placebo (Placebo Comparator): Participants receive frespaciguat-matching placebo QD via inhalation from Days 1-7.
  Interventions: Drug: Placebo
- Panel B Frespaciguat 360 µg (Experimental): Participants receive 360 µg of frespaciguat QD via inhalation from Days 1-7.
  Interventions: Drug: Frespaciguat
- Panel B Placebo (Placebo Comparator): Participants receive frespaciguat-matching placebo QD via inhalation from Days 1-7.
  Interventions: Drug: Placebo
- Panel C Frespaciguat ≤360 µg (Experimental): Participants receive ≤360 µg of frespaciguat QD via inhalation from Days 1-7.
  Interventions: Drug: Frespaciguat
- Panel C Placebo (Placebo Comparator): Participants receive frespaciguat-matching placebo QD via inhalation from Days 1-7.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Frespaciguat — Frespaciguat administered at a dose of 180 µg or ≤360 µg QD via inhalation
  Other Names: MK-5475
  Arms: Panel A Frespaciguat 180 µg; Panel B Frespaciguat 360 µg; Panel C Frespaciguat ≤360 µg
Drug: Placebo — Frespaciguat-matching placebo administered QD via inhalation
  Arms: Panel A Placebo; Panel B Placebo; Panel C Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, and pharmacodynamics of frespaciguat after administration of multiple doses to participants with COVID-19 pneumonia. The primary hypothesis is that frespaciguat when administered to participants with COVID-19 pneumonia and hypoxemia improves arterial oxygenation as measured by the ratio of blood oxygen saturation to fraction of inspired oxygen (SpO2/FiO2 ratio) compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Has virologically confirmed COVID-19 requiring hospital admission.
* Has respiratory symptoms including cough and dyspnea
* Requires supplemental oxygen therapy
* Male participant is abstinent from heterosexual intercourse or agrees to use contraception during the intervention period and for at least 14 days, corresponding to time needed to eliminate study intervention(s) (example, 5 terminal half-lives after the last dose of study intervention)
* Female participant is not a woman of childbearing potential (WOCBP) or is a WOCBP who is abstinent from heterosexual intercourse or using contraception during the intervention period and for at least 14 days, corresponding to time needed to eliminate study intervention(s) (example, 5 terminal half-lives after the last dose of study intervention)

Exclusion Criteria:

* Has pre-existing medical conditions of any nature which are immediately pre-terminal such as death or limitation of life-sustaining therapy is expected to be imminent
* Requires or is expected to require invasive mechanical ventilation
* Requires or is expected to require noninvasive mechanical ventilation
* Has any issue which would prohibit them from effective use of the frespaciguat inhaler
* Hypoxemia which is explained by any condition other than COVID-19, example, preexisting cardiac or pulmonary disease
* Has severe hepatic impairment (meets Child-Pugh Class C criteria)
* Has severe renal impairment and/or requirement for renal dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-07 (Estimated); Primary Completion 2020-11-10 (Estimated); Study Completion 2020-11-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to ~Day 21
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinued Study Drug Due to an Adverse Event (AE) | Up to ~Day 7
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study drug due to an AE will be reported.
Change From Baseline to Day 1 in the Time-weighted Average from 0 through 24 hours (TWA0-24hrs) for the Ratio of Blood Oxygen Saturation to the Fraction of Inspired Oxygen (SpO2/FiO2) | Baseline, Day 1 (pre-dose and 2, 6, 12, 18, 24 hours post-dose)
  The SpO2/FiO2 ratio is a measure of arterial oxygenation. Noninvasive pulse oximetry will be used to obtain the SpO2/FiO2 ratio. The TWA0-24hrs will be calculated as the area under the curve from 0 to 24 hours post-dose on Day 1 divided by the length of time (24 hrs). Baseline is the Day 1 pre-dose measurement and assessments will be conducted pre-dose and at multiple time points post-dose on Day 1 to determine change from baseline in TWA0-24hrs for SpO2/FiO2 on Day 1.
Change From Baseline to Day 2 in the Time-weighted Average from 0 through 24 hours (TWA0-24hrs) for the Ratio of Blood Oxygen Saturation to the Fraction of Inspired Oxygen (SpO2/FiO2) | Baseline, Day 2 (pre-dose and 2, 6, 12, 18, 24 hours post-dose)
  The SpO2/FiO2 ratio is a measure of arterial oxygenation. Noninvasive pulse oximetry will be used to obtain the SpO2/FiO2 ratio. The TWA0-24hrs will be calculated as the area under the curve from 0 to 24 hours on Day 2 divided by the length of time (24 hrs). Baseline is the Day 1 pre-dose measurement and assessments will be conducted pre-dose and at multiple time points post-dose on Day 2 to determine change from baseline in TWA0-24hrs for SpO2/FiO2 on Day 2.
Change From Baseline to Day 3 in the Time-weighted Average from 0 through 24 hours (TWA0-24hrs) for the Ratio of Blood Oxygen Saturation to the Fraction of Inspired Oxygen (SpO2/FiO2) | Baseline, Day 3 (pre-dose and 2, 6, 12, 18, 24 hours post-dose)
  The SpO2/FiO2 ratio is a measure of arterial oxygenation. Noninvasive pulse oximetry will be used to obtain the SpO2/FiO2 ratio. The TWA0-24hrs will be calculated as the area under the curve from 0 to 24 hours on Day 3 divided by the length of time (24 hrs). Baseline is the Day 1 pre-dose measurement and assessments will be conducted pre-dose and at multiple time points post-dose on Day 3 to determine change from baseline in TWA0-24hrs for SpO2/FiO2 on Day 3.
Change From Baseline to Day 4 in the Time-weighted Average from 0 through 24 hours (TWA0-24hrs) for the Ratio of Blood Oxygen Saturation to the Fraction of Inspired Oxygen (SpO2/FiO2) | Baseline, Day 4 (pre-dose and 2, 6, 12, 18, 24 hours post-dose)
  The SpO2/FiO2 ratio is a measure of arterial oxygenation. Noninvasive pulse oximetry will be used to obtain the SpO2/FiO2 ratio. The TWA0-24hrs will be calculated as the area under the curve from 0 to 24 hours on Day 4 divided by the length of time (24 hrs). Baseline is the Day 1 pre-dose measurement and assessments will be conducted pre-dose and at multiple time points post-dose on Day 4 to determine change from baseline in TWA0-24hrs for SpO2/FiO2 on Day 4.
Change From Baseline to Day 5 in the Time-weighted Average from 0 through 24 hours (TWA0-24hrs) for the Ratio of Blood Oxygen Saturation to the Fraction of Inspired Oxygen (SpO2/FiO2) | Baseline, Day 5 (pre-dose and 2, 6, 12, 18, 24 hours post-dose)
  The SpO2/FiO2 ratio is a measure of arterial oxygenation. Noninvasive pulse oximetry will be used to obtain the SpO2/FiO2 ratio. The TWA0-24hrs will be calculated as the area under the curve from 0 to 24 hours on Day 5 divided by the length of time (24 hrs). Baseline is the Day 1 pre-dose measurement and assessments will be conducted pre-dose and at multiple time points post-dose on Day 5 to determine change from baseline in TWA0-24hrs for SpO2/FiO2 on Day 5.
Change From Baseline to Day 6 in the Time-weighted Average from 0 through 24 hours (TWA0-24hrs) for the Ratio of Blood Oxygen Saturation to the Fraction of Inspired Oxygen (SpO2/FiO2) | Baseline, Day 6 (pre-dose and 2, 6, 12, 18, 24 hours post-dose)
  The SpO2/FiO2 ratio is a measure of arterial oxygenation. Noninvasive pulse oximetry will be used to obtain the SpO2/FiO2 ratio. The TWA0-24hrs will be calculated as the area under the curve from 0 to 24 hours on Day 6 divided by the length of time (24 hrs). Baseline is the Day 1 pre-dose measurement and assessments will be conducted pre-dose and at multiple time points post-dose on Day 6 to determine change from baseline in TWA0-24hrs for SpO2/FiO2 on Day 6.
Change From Baseline to Day 7 in the Time-weighted Average from 0 through 24 hours (TWA0-24hrs) for the Ratio of Blood Oxygen Saturation to the Fraction of Inspired Oxygen (SpO2/FiO2) | Baseline, Day 7 (pre-dose and 2, 6, 12, 18, 24 hours post-dose)
  The SpO2/FiO2 ratio is a measure of arterial oxygenation. Noninvasive pulse oximetry will be used to obtain the SpO2/FiO2 ratio. The TWA0-24hrs will be calculated as the area under the curve from 0 to 24 hours on Day 7 divided by the length of time (24 hrs). Baseline is the Day 1 pre-dose measurement and assessments will be conducted pre-dose and at multiple time points post-dose on Day 7 to determine change from baseline in TWA0-24hrs for SpO2/FiO2 on Day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/